CLINICAL TRIAL: NCT06845904
Title: Study on Preliminary Safety and Efficacy of Epidural Electrical Stimulation to Manage Lower Urinary Tract Dysfunction After Spinal Cord Injury
Acronym: ReeVoid
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ecole Polytechnique Fédérale de Lausanne (Other)
Responsible Party: Principal Investigator, Jocelyne Bloch, Prof., Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ReeVoid
Record Dates: First submitted 2025-01-28; First posted 2025-02-25 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Spinal Cord Injuries (SCI); Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Single-site, single-arm, non-blinded, non-randomized, interventional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): All participants enrolled in the study will receive the same intervention. This clinical trial evaluates a novel therapy using a CE-marked medical device employed off-label. Participants will undergo implantation of a neurostimulation system designed to deliver electrical stimulation to the spinal cord. The therapy aims to improve control over detrusor and urethral sphincter muscles by targeting the associated nerves.
  Interventions: Device: WaveWriter Alpha™ neurostimulation system

INTERVENTIONS:
Device: WaveWriter Alpha™ neurostimulation system — Two Boston Scientific WaveWriter Alpha™ Implantable Pulse Generators (IPGs) will be implanted and connected to CoverEdge™ or CoverEdge™ X 32 Surgical Paddle Leads. The leads are positioned to enable targeted stimulation of the spinal cord to optimize control of urinary functions.

SUMMARY:
This clinical trial aims to assess the preliminary safety and efficacy of Epidural Electrical Stimulation (EES) therapy in managing lower urinary tract dysfunction in individuals with sub-acute or chronic spinal cord injury (SCI). The study evaluates the therapy's potential to improve urinary function and prevent neurogenic detrusor overactivity, ultimately seeking to enhance quality of life for individuals with SCI.

DETAILED DESCRIPTION:
The consequences of a Spinal Cord Injury (SCI) are dramatic. SCI leads to impairment of motor, sensory, and autonomic systems, dysregulating almost every bodily function below the level of injury. The majority of research on SCI focuses on the restoration of movement. However, the disruption of pathways controlling the bladder leads to less-appreciated symptoms that require life-long clinical management, are the one of the main cause of rehospitalization, and incurred the largest healthcare costs after SCI. Neurogenic bladder issues, such as neurogenic detrusor overactivity (NDO) leading to incontinence, detrusor-sphincter dyssynergia (DSD) and decreased bladder compliance, are currently treated with intermittent catheterization, anticholinergic medications, botulinum toxin injections directly into the detrusor and ultimately irreversible major surgical interventions. Despite improvement in bladder management provided by these clinical and interventional tools, people with SCI still experience recurrent urinary tract infections from repeated catheterization, incontinence events impacting their professional and intimate life, side-effects from anti-cholinergic medication. It therefore comes as no surprise that people with spinal cord injury prioritize the treatment of lower urinary tract dysfunction as one of their top health priorities.

The investigators reasoned that the neuroprosthetic management of micturition and urinary continence may overcome many of the existing limitations of current clinical management strategies. To test this idea, the investigators have developed a neuroprosthetic system based on Epidural Electrical Stimulation (EES) of the spinal cord that restored micturition (EESVOIDING) and improve urinary continence by reducing detrusor overactivity (EESSTORAGE) in preclinical models of SCI. Development of this neuroprosthetic system combined with rigorous experiments led to the identification of the locations and parameters of EES that can activate the detrusor while relaxing the external urethral sphincter (EUS). The investigators also gathered preliminary evidence on the key features of this therapeutic strategy in one patient with low-thoracic motor-complete SCI (T10, AIS-B) who was implanted with a neuroprosthetic system on the lumbosacral spinal cord (covering T12 to S1) to restore walking (STIMO clinical Trial, NCT02936453). Stimulation of the sacral spinal cord of this participant resulted in controlled detrusor contraction leading to voiding. Consequently, the investigators hypothesize that EES has the potential to become the first-line treatment for bladder dysfunction in people with chronic or sub-acute SCI. However, its clinical deployment relies on selective stimulation paradigms and development of medical-grade implantable spinal-cord stimulation technologies that are optimized for bladder management.

The ReeVoid clinical study will enroll 3 participants, who will be implanted with a system to apply EES to stimulate the spinal circuits involved in the control of the bladder. The aim of the study is to manage lower urinary tract functions with EES, including supporting voiding and preventing neurogenic detrusor overactivity incontinence (NDOI) in individuals with sub-acute or chronic spinal cord injury located above T11 and who suffer from lower urinary tract dysfunction. Two electrode paddle leads will be implanted. The first one will cover the dorsal root entry zone of the lumbosacral segments (L4-S5), while the second will aim to target the S1-S4 roots where they exit the spinal canal in the lower vertebras, and thus to maximise selective recruitment of the dorsal roots involved in the control of the detrusor and urethral sphincter muscles. Each paddle lead will be connected to a neurostimulator located subcutaneously in the region of the abdomen.

This therapy aims also to have a positive impact on other neurological functions such as sexual function, bowel management and muscle tone normalization (reduced spasticity).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older;
* Must provide and sign the Informed Consent Form prior to any study-related procedures;
* Spinal cord injury lesion level above T11 (inclusive);
* SCI graded as AIS- B, C or D;
* SCI ≥ 6 months;
* Confirmed lower urinary tract dysfunction during urodynamic assessment (NDO, DSD);
* Intolerant, refractory or inefficient to conservative treatment options such as medications and behavioural management;
* Using intermittent self-catheterization;
* Stable medical, physical and psychological condition as considered by the investigators;
* Able to understand and interact with the study team in French or English;
* Agrees to comply in good faith with all conditions of the study and to attend all scheduled appointments;

Exclusion Criteria:

* Botulinum toxin vesical injections in the previous 6 months;
* Presence of non-pharmacological treatments for lower urinary tract dysfunction (e.g. sacral nerve stimulation);
* Does have or needs a suprapubic catheter or bladder indwelling catheter;
* Presence of upper urinary tract dilatation or bladder or renal stones;
* Presence of urethral stricture or significant benign prostate hyperplasia;
* Presence of significant pressure ulcers;
* Previous lower urinary tract surgery;
* Presence of Autonomic Dysreflexia during urodynamic test;
* Recurrent and symptomatic urinary tract infection (more than 3 per year);
* Presence of intrathecal baclofen pump;
* Diseases and conditions that would increase the morbidity and mortality of spinal surgery;
* Other clinically significant concomitant disease states (e.g., syringomyelia, bladder cancer, renal failure, hepatic dysfunction, cardiovascular disease, etc.);
* The inability to withhold antiplatelet/anticoagulation agents perioperatively;
* Presence of pacemakers for cardiac conditions;
* Other conditions that would make the subject unable to participate in testing in the judgement of the investigators;
* Women who are pregnant (pregnancy test obligatory for woman of childbearing potential) or breast feeding;
* Lack of acceptable or highly effective method of contraception for women of childbearing capacity;
* Intention to become pregnant during the course of the study;
* Inability to follow the procedures of the study, e.g. due to language problems, mental illness, psychological disorders, or dementia of the participant;
* Participation in another study with investigational drug or device within the 30 days preceding and during the present study;
* Have any indication that would require Magnetic Resonance Imaging (MRI)
* Is the investigator himself, his/her family members, employees or other dependent persons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Occurrence of serious adverse events and adverse events. | From enrolment through study completion, an average of 10 months.
  Occurrence of serious adverse events and adverse events that are deemed related or possibly related to the use of the investigational.

SECONDARY OUTCOMES:
ASIA impairment scale - International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) | Pre-implantation (up to 3 weeks pre-implantation) and at the End of Study phase (lasting up to 1 week at 9 months)
  Clinical examination used to assess the motor and sensory impairment and severity of a spinal cord injury.
Spasticity assessment (Modified Ashworth Scale - MAS) | Pre-implantation (up to 2 weeks pre-implantation) and at Follow-up phase and End of Study phase (at months 3, 6 and 9 post-implantation and lasting up to 1 week)
  Resistance of a muscle to a passive range of motion about a single joint, measured using the Modified Ashworth Scale (MAS), a 6-point scale with scores of 0, 1, 1+, 2, 3, and 4. A score of 0 indicates no increase in muscle tone, while a score of 4 indicates the affected part is rigid in flexion or extension. Higher scores indicate worse spasticity.
Daily Bladder related diary | Pre-implantation (up to 2 weeks pre-implantation), Mapping phase (1 week post-implantation and lasting up to 1 month), at Follow-up phase and End of Study phase (at months 3 and 6 post-implantation and lasting up to 1 week)
  Self-reported measures including urinary related events (voiding volume by catheterization and electrical stimulation, frequency, daytime and during night frequency, catheterization and volume of residual volume after stimulation, symptomatic urinary tract infection, use of stimulation) reported on a tracking app to quantify changes before and after implantation.
Renal ultrasound | Pre-implantation (up to 3 weeks before implantation), Mapping phase (1 week post-implantation and lasting up to 1 month), Follow-up phase and End of Study phase (at months 3, 6 and 9 post-implantation and lasting up to 1 week)
  Renal ultrasound is used to monitor the kidneys, ureters, and bladder, providing valuable information about kidney size, shape, and position.
Urine sampling | Pre-implantation (up to 3 weeks pre-implantation) and upon suspicion
  Urine sampling is taken to confirm the absence of any urinary tract.
24 hours urine collection | Pre-implantation (up to 3 weeks pre-implantation) and at Follow-up phase and End of Study phase (at months 3, 6 and 9 post-implantation and lasting up to 1 week)
  24 hours urine collection is taken to quantify the spot albumin and creatinine in the urine. These parameters are used to confirm the absence of any renal dysfunctions.
Blood samples | Pre-implantation (up to 3 weeks pre-implantation) and at Follow-up phase and End of Study phase (at months 3, 6 and 9 post-implantation and lasting up to 1 week)
  Blood sampling (max 20mL) is taken to quantify creatinine, aspartate aminotransferase (AST), alanine aminotransferase (ALT) and cystatin C. These parameters are used to confirm the absence of any renal dysfunctions.
Cystometry | Pre-implantation (up to 3 weeks and up to 2 weeks pre-implantation), Mapping phase (1 week post-implantation and lasting up to 1 month), at Follow-up phase and End of Study phase (at months 3, 6 and 9 post-implantation and lasting up to 1 week)
  A catheter is inserted into the bladder to measure intravesical pressure while the bladder is filled with sterile fluid at a controlled rate. Simultaneously, abdominal pressure is monitored to assess detrusor pressure and bladder compliance. Cystometry helps identify neurogenic detrusor overactivity, bladder capacity, and compliance.
Imaging (with contrast agent) | Pre-implantation (up to 3 weeks and up to 2 weeks pre-implantation), Mapping phase (1 week post-implantation and lasting up to 1 month), at Follow-up phase and End of Study phase (at months 3, 6 and 9 post-implantation and lasting up to 1 week)
  X-Ray (or fluoroscopy) can be taken, with imaging contrast agents, to provide visualization of the urinary tract and/or catheter placements (optional).
Pressure-flow study | Pre-implantation (up to 3 weeks and up to 2 weeks pre-implantation), Mapping phase (1 week post-implantation and lasting up to 1 month), at Follow-up phase and End of Study phase (at months 3, 6 and 9 post-implantation and lasting up to 1 week)
  During voiding, simultaneous measurements of detrusor pressure and urinary flow rate are recorded. This aids in diagnosing detrusor-sphincter dyssynergia (DSD), evaluating voiding efficiency, and identifying obstructive patterns.
Electromyography (EMG) | Pre-implantation (up to 3 weeks and up to 2 weeks pre-implantation), Mapping phase (1 week post-implantation and lasting up to 1 month), at Follow-up phase and End of Study phase (at months 3, 6 and 9 post-implantation and lasting up to 1 week)
  Surface electrodes or specialized catheters are used to record electrical activity in the bladder and external urethral sphincter muscles. EMG helps detect detrusor-sphincter dyssynergia (DSD) by assessing the coordination between detrusor and sphincter activity during filling and voiding.
Flowmetry - Urethral pressure profile (UPP) | Pre-implantation (up to 3 weeks and up to 2 weeks pre-implantation), Mapping phase (1 week post-implantation and lasting up to 1 month), at Follow-up phase and End of Study phase (at months 3, 6 and 9 post-implantation and lasting up to 1 week)
  A catheter-mounted pressure sensor is withdrawn slowly from the bladder through the urethra, recording pressure changes along the urethral length. UPP assists in evaluating sphincter function and diagnosing urethral obstruction.

OTHER OUTCOMES:
NBDS (Neurogenic Bowel Dysfunction Score) | Pre-implantation (up to 2 weeks pre-implantation) and monthly for 9 months post-implantation
  10-item questionnaire that is associated with impaired QoL caused by bowel symptoms. The NBD weighted score ranges between 0 and 47 points. A higher overall NBD score indicates more severe bowel symptoms.
NBSS (Neurogenic Bladder Symptom Score) | Pre-implantation (up to 2 weeks pre-implantation) and monthly for 9 months post-implantation
  The NBSS consists of 24 items across three domains: Incontinence (scored 0-29); Storage and Voiding (scored 0-22); and Consequences (scored 0-23). For all domains, a higher score represents a worse symptom burden or QoL (quality of life).
SF-Qualiveen (QUALIVEEN Short Form) | Pre-implantation (up to 2 weeks pre-implantation) and monthly for 9 months post-implantation
  To assess health-related quality of life of patients with urinary disorders in neurologic conditions. The 8-item questionnaire include bother with limitations (2 items), frequency of limitations (2 items), fears (2 items), and feelings (2 items). Items 1-6 are scored on a 5-point scale (0 to 4), with higher scores indicating a greater negative impact on quality of life. Items 7-8 are scored on a 5-point reverse scale (0 to 4), where higher scores indicate less impact on quality of life.
IIEF/FSFI (International Index of Erectile Function-5/Female Sexual Function Index) | Pre-implantation (up to 2 weeks pre-implantation) and monthly for 9 months post-implantation
  IIEF-15: A 15-item questionnaire covering five domains: erectile function (6 items), orgasmic function (2 items), sexual desire (2 items), intercourse satisfaction (3 items), and overall satisfaction (2 items). Scores range from 5 to 25, with erectile dysfunction (ED) classified as severe (5-7), moderate (8-11), mild to moderate (12-16), mild (17-21), and no ED (22-25). Higher scores indicate better erectile function.
  FSFI: A 19-item self-reported measure assessing six domains: desire, subjective arousal, lubrication, orgasm, satisfaction, and pain. Each item is scored on a 5-point scale (1 to 5), with higher scores indicating better sexual function.
ADFSCI (Autonomic Dysreflexia following SCI) | Pre-implantation (up to 3 weeks pre-implantation) and monthly for 9 months post-implantation
  The ADFSCI is a 24-item questionnaire consisting of four parts: demographics, medication, AD (Autonomic Dysreflexia) and hypotension. The AD section (10 items) and hypotension section (7 items) assess the severity and frequency of hyper- or hypotensive symptoms, such as headache, goosebumps, dizziness, and light-headedness, in different circumstances. Each item is scored on a 5-point scale (0 to 4), with higher scores indicating greater severity and frequency of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyne Bloch, MD, Principal Investigator — Centre hospitalier universitaire vaudois (CHUV)
Locations (1):
- Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perrouin-Verbe B, Labat JJ, Richard I, Mauduyt de la Greve I, Buzelin JM, Mathe JF. Clean intermittent catheterisation from the acute period in spinal cord injury patients. Long term evaluation of urethral and genital tolerance. Paraplegia. 1995 Nov;33(11):619-24. doi: 10.1038/sc.1995.131. PMID 8584294
- [Background] Harkema S, Gerasimenko Y, Hodes J, Burdick J, Angeli C, Chen Y, Ferreira C, Willhite A, Rejc E, Grossman RG, Edgerton VR. Effect of epidural stimulation of the lumbosacral spinal cord on voluntary movement, standing, and assisted stepping after motor complete paraplegia: a case study. Lancet. 2011 Jun 4;377(9781):1938-47. doi: 10.1016/S0140-6736(11)60547-3. Epub 2011 May 19. PMID 21601270
- [Background] Herrity AN, Williams CS, Angeli CA, Harkema SJ, Hubscher CH. Lumbosacral spinal cord epidural stimulation improves voiding function after human spinal cord injury. Sci Rep. 2018 Jun 6;8(1):8688. doi: 10.1038/s41598-018-26602-2. PMID 29875362
- [Background] Walter M, Lee AHX, Kavanagh A, Phillips AA, Krassioukov AV. Epidural Spinal Cord Stimulation Acutely Modulates Lower Urinary Tract and Bowel Function Following Spinal Cord Injury: A Case Report. Front Physiol. 2018 Dec 18;9:1816. doi: 10.3389/fphys.2018.01816. eCollection 2018. PMID 30618826
- [Background] Rowald A, Komi S, Demesmaeker R, Baaklini E, Hernandez-Charpak SD, Paoles E, Montanaro H, Cassara A, Becce F, Lloyd B, Newton T, Ravier J, Kinany N, D'Ercole M, Paley A, Hankov N, Varescon C, McCracken L, Vat M, Caban M, Watrin A, Jacquet C, Bole-Feysot L, Harte C, Lorach H, Galvez A, Tschopp M, Herrmann N, Wacker M, Geernaert L, Fodor I, Radevich V, Van Den Keybus K, Eberle G, Pralong E, Roulet M, Ledoux JB, Fornari E, Mandija S, Mattera L, Martuzzi R, Nazarian B, Benkler S, Callegari S, Greiner N, Fuhrer B, Froeling M, Buse N, Denison T, Buschman R, Wende C, Ganty D, Bakker J, Delattre V, Lambert H, Minassian K, van den Berg CAT, Kavounoudias A, Micera S, Van De Ville D, Barraud Q, Kurt E, Kuster N, Neufeld E, Capogrosso M, Asboth L, Wagner FB, Bloch J, Courtine G. Activity-dependent spinal cord neuromodulation rapidly restores trunk and leg motor functions after complete paralysis. Nat Med. 2022 Feb;28(2):260-271. doi: 10.1038/s41591-021-01663-5. Epub 2022 Feb 7. PMID 35132264
- [Background] Jantz MK, Gopinath C, Kumar R, Chin C, Wong L, Ogren JI, Fisher LE, McLaughlin BL, Gaunt RA. High-density spinal cord stimulation selectively activates lower urinary tract nerves. J Neural Eng. 2022 Nov 22;19(6):066014. doi: 10.1088/1741-2552/aca0c2. PMID 36343359
- [Background] Squair JW, Gautier M, Mahe L, Soriano JE, Rowald A, Bichat A, Cho N, Anderson MA, James ND, Gandar J, Incognito AV, Schiavone G, Sarafis ZK, Laskaratos A, Bartholdi K, Demesmaeker R, Komi S, Moerman C, Vaseghi B, Scott B, Rosentreter R, Kathe C, Ravier J, McCracken L, Kang X, Vachicouras N, Fallegger F, Jelescu I, Cheng Y, Li Q, Buschman R, Buse N, Denison T, Dukelow S, Charbonneau R, Rigby I, Boyd SK, Millar PJ, Moraud EM, Capogrosso M, Wagner FB, Barraud Q, Bezard E, Lacour SP, Bloch J, Courtine G, Phillips AA. Neuroprosthetic baroreflex controls haemodynamics after spinal cord injury. Nature. 2021 Feb;590(7845):308-314. doi: 10.1038/s41586-020-03180-w. Epub 2021 Jan 27. PMID 33505019
- [Background] Soriano JE, Squair JW, Cragg JJ, Thompson J, Sanguinetti R, Vaseghi B, Emery CA, Grant C, Charbonneau R, Larkin-Kaiser KA, Phillips AA, Dujic Z. A national survey of physical activity after spinal cord injury. Sci Rep. 2022 Mar 15;12(1):4405. doi: 10.1038/s41598-022-07927-5. PMID 35292668
- [Background] Hoey RF, Medina-Aguinaga D, Khalifa F, Ugiliweneza B, Zdunowski S, Fell J, Naglah A, El-Baz AS, Herrity AN, Harkema SJ, Hubscher CH. Bladder and bowel responses to lumbosacral epidural stimulation in uninjured and transected anesthetized rats. Sci Rep. 2021 Feb 8;11(1):3268. doi: 10.1038/s41598-021-81822-3. PMID 33558526
- [Background] Herrity AN, Aslan SC, Mesbah S, Siu R, Kalvakuri K, Ugiliweneza B, Mohamed A, Hubscher CH, Harkema SJ. Targeting bladder function with network-specific epidural stimulation after chronic spinal cord injury. Sci Rep. 2022 Jul 1;12(1):11179. doi: 10.1038/s41598-022-15315-2. PMID 35778466
- [Background] Wagner FB, Mignardot JB, Le Goff-Mignardot CG, Demesmaeker R, Komi S, Capogrosso M, Rowald A, Seanez I, Caban M, Pirondini E, Vat M, McCracken LA, Heimgartner R, Fodor I, Watrin A, Seguin P, Paoles E, Van Den Keybus K, Eberle G, Schurch B, Pralong E, Becce F, Prior J, Buse N, Buschman R, Neufeld E, Kuster N, Carda S, von Zitzewitz J, Delattre V, Denison T, Lambert H, Minassian K, Bloch J, Courtine G. Targeted neurotechnology restores walking in humans with spinal cord injury. Nature. 2018 Nov;563(7729):65-71. doi: 10.1038/s41586-018-0649-2. Epub 2018 Oct 31. PMID 30382197
- [Background] Kathe C, Skinnider MA, Hutson TH, Regazzi N, Gautier M, Demesmaeker R, Komi S, Ceto S, James ND, Cho N, Baud L, Galan K, Matson KJE, Rowald A, Kim K, Wang R, Minassian K, Prior JO, Asboth L, Barraud Q, Lacour SP, Levine AJ, Wagner F, Bloch J, Squair JW, Courtine G. The neurons that restore walking after paralysis. Nature. 2022 Nov;611(7936):540-547. doi: 10.1038/s41586-022-05385-7. Epub 2022 Nov 9. PMID 36352232
- [Background] Anderson MA, Squair JW, Gautier M, Hutson TH, Kathe C, Barraud Q, Bloch J, Courtine G. Natural and targeted circuit reorganization after spinal cord injury. Nat Neurosci. 2022 Dec;25(12):1584-1596. doi: 10.1038/s41593-022-01196-1. Epub 2022 Nov 17. PMID 36396975
- [Background] McGee MJ, Amundsen CL, Grill WM. Electrical stimulation for the treatment of lower urinary tract dysfunction after spinal cord injury. J Spinal Cord Med. 2015 Mar;38(2):135-46. doi: 10.1179/2045772314Y.0000000299. Epub 2015 Jan 13. PMID 25582564
- [Background] Groenendijk IM, Groen J, Scheepe JR, Blok BFM. Acute effect of sacral neuromodulation for treatment of detrusor overactivity on urodynamic parameters. Neurourol Urodyn. 2020 Feb;39(2):695-701. doi: 10.1002/nau.24252. Epub 2019 Dec 5. PMID 31804759
- [Background] Capogrosso M, Wenger N, Raspopovic S, Musienko P, Beauparlant J, Bassi Luciani L, Courtine G, Micera S. A computational model for epidural electrical stimulation of spinal sensorimotor circuits. J Neurosci. 2013 Dec 4;33(49):19326-40. doi: 10.1523/JNEUROSCI.1688-13.2013. PMID 24305828
- [Background] Squair JW, Dhaliwal R, Cragg JJ, Charbonneau R, Grant C, Phillips AA. National Survey of Bladder and Gastrointestinal Dysfunction in People with Spinal Cord Injury. J Neurotrauma. 2019 Jun 15;36(12):2011-2019. doi: 10.1089/neu.2018.5967. Epub 2019 Jan 25. PMID 30501555
- [Background] Panicker JN, Fowler CJ, Kessler TM. Lower urinary tract dysfunction in the neurological patient: clinical assessment and management. Lancet Neurol. 2015 Jul;14(7):720-32. doi: 10.1016/S1474-4422(15)00070-8. PMID 26067125
- [Background] Hou S, Rabchevsky AG. Autonomic consequences of spinal cord injury. Compr Physiol. 2014 Oct;4(4):1419-53. doi: 10.1002/cphy.c130045. PMID 25428850
- [Background] Ackery A, Tator C, Krassioukov A. A global perspective on spinal cord injury epidemiology. J Neurotrauma. 2004 Oct;21(10):1355-70. doi: 10.1089/neu.2004.21.1355. PMID 15672627